CLINICAL TRIAL: NCT02753894
Title: Phase II Dose Range-finding Study of ASP1585 in Chronic Kidney Disease Patients on Hemodialysis With Hyperphosphatemia
Brief Title: Dose Range-finding Study of ASP1585 in Chronic Kidney Disease Patients on Hemodialysis With Hyperphosphatemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1585-CL-0006
Record Dates: First submitted 2016-03-03; First posted 2016-04-28 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Kidney Disease Patients on Hemodialysis With Hyperphosphatemia
Keywords: Dose-finding; Hemodialysis; ASP1585; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — bixalomer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4.5 g/day group (Experimental): Three times a day
  Interventions: Drug: ASP1585
- 6.0 g/day group (Experimental): Three times a day
  Interventions: Drug: ASP1585
- 7.5 g/day group (Experimental): Three times a day
  Interventions: Drug: ASP1585

INTERVENTIONS:
Drug: ASP1585 — Oral
  Other Names: Bixalomer; Kiklin (R)

SUMMARY:
The objective of this study is to examine the clinical dose range of ASP1585 based on the efficacy, safety, and feasibility of treatment in chronic kidney disease patients on hemodialysis with hyperphosphatemia.

ELIGIBILITY:
Inclusion Criteria:

For preliminary enrollment

* Patients with stable chronic kidney disease who received hemodialysis 3 times a week for at least 12 weeks (84 days) prior to the day of preliminary enrollment
* Patients who did not have dialysis conditions altered (dialysate calcium concentration, dialyser, and dry weight) within 10 days prior to the day of preliminary enrollment
* Patients who did not have the following dosage or administration altered at least 28 days prior to the day of preliminary enrollment: phosphate binders, or drugs/food with phosphate binding action (including newly started treatment)
* If receiving vitamin D or calcitonin agent, patients who did not have dosage and administration altered (including newly started treatment) for at least 28 days prior to the day of preliminary enrollment.
* Patients who did not use cinacalcet hydrochloride for at least 28 days prior to the day of preliminary enrollment

For practical enrollment

* Patients whose pre-dialysis serum phosphorus level after the maximum dialysis interval at Week 1 of the washout period was ≥8.0 mg/dL and <10.0 mg/dL or that at Week 2 was ≥6.0 mg/dL and <10.0 mg/dL
* Patients who continued to receive hemodialysis 3 times a week after the day of preliminary enrollment
* Patients who did not have dialysis conditions altered (dialysate calcium concentration and dialyser) after the day of preliminary enrollment
* Patients who did not receive phosphate binders, or drugs/food with phosphate binding action during the washout period
* If receiving vitamin D or calcitonin agent (including start of new treatment) after the day of preliminary enrollment, patients who did not have dosage and administration altered for at least 28 days prior to the day of preliminary enrollment
* Patients who did not use cinacalcet hydrochloride after the day of preliminary enrollment

Exclusion Criteria:

For preliminary enrollment

* Patients with a history of gastrectomy or enterectomy (except for appendectomy) or with a complication of dysphagia, ileus, or hemorrhagic gastrointestinal lesions
* Patients with severe persistent constipation or diarrhoea
* Patients who underwent parathyroid intervention (parathyroidectomy [PTx], percutaneous ethanol injection therapy [PEIT], etc.) within 1 year prior to the day of preliminary enrollment
* Patients who are fasted or are on extreme dietary restrictions
* Patients with uncontrollable hypertension (all the last 3 measurement values of pre-dialysis systolic/diastolic blood pressure before the day of preliminary enrollment are ≥180 mmHg and ≥120 mmHg, respectively)
* Patients with severe heart disease (congestive heart failure [NYHA cardiac function classification Class III or severer], a history of extensive old myocardial infarction, etc.) or patients who were hospitalized for the treatment of cerebrovascular disease or heart disease within 12 weeks (84 days) prior to the day of preliminary enrollment
* Patients with a complication of serious hepatic disease (acute and active chronic hepatitis, hepatic cirrhosis, etc.)
* Patients with a history of serious drug hypersensitivity, such as anaphylactic shock
* Patients with a history or complication of malignant tumor (considered eligible if recurrence has not been observed for at least 5 years)
* Patients who are pregnant, nursing, suspected to be pregnant, or wish to become pregnant during the study period
* Patients who have previously received ASP1585
* Patients who participated in another clinical study or a post-marketing clinical study (including that of a medical device) within 12 weeks (84 days) prior to informed consent

For practical enrollment

* Patients whose pre-dialysis serum phosphorus level after the maximum dialysis interval at Week 1 or 2 of the washout period was ≥10 mg/dL
* Patients who underwent gastrectomy or enterectomy, or had dysphagia, ileus, or hemorrhagic gastrointestinal lesions after the day of preliminary enrollment
* Patents who had severe persistent constipation or diarrhoea after the day of preliminary enrollment
* Patients who underwent parathyroid intervention (parathyroidectomy [PTx], percutaneous ethanol injection therapy [PEIT], etc.) after the day of preliminary enrollment
* Patients who were fasted or on extreme dietary restriction after the day of preliminary enrollment
* Patients with uncontrollable hypertension (more than two thirds of pre-dialysis systolic/diastolic blood pressure values were ≥180 mmHg and ≥120 mmHg, respectively, after the day of preliminary enrollment)
* Patients with severe heart disease (congestive heart failure [NYHA cardiac function classification Class III or severer], etc.) or patients who were hospitalized for the treatment of cerebrovascular disease or heart disease after the day of preliminary enrollment
* Patients with a complication of impaired liver function (baseline AST or ALT was 100 IU/L or higher) or serious hepatic disease (acute and active chronic hepatitis, liver cirrhosis, etc.)
* Patients who experienced serious drug hypersensitivity such as anaphylactic shock after the day of preliminary enrollment
* Patients with a complication of malignant tumor
* Patients who were found to be pregnant after the day of preliminary enrollment
* Patients who participated in another clinical study or a post-marketing clinical study (including that of a medical device) after the day of informed consent

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change from the baseline of serum phosphorus level | Baseline and Week 6
Safety assessed by AEs | Up to 6 weeks after the study drug dosing
Safety assessed by Hematology test | Up to 6 weeks after the study drug dosing
Safety assessed by Blood biochemistry tests | Up to 6 weeks after the study drug dosing
Safety assessed by Blood cogulability tests | Up to 6 weeks after the study drug dosing
Blood concentration of Vitamin | Up to 6 weeks after the study drug dosing
Safety assessed by Vital signs | Up to 6 weeks after the study drug dosing
  Systolic blood pressure, diastolic blood pressure, heart rate
Safety assessed by bowel movement | Up to 6 weeks after the study drug dosing
Safety assessed by ECG | Up to 6 weeks after the study drug dosing

SECONDARY OUTCOMES:
Time course of serum phosphorus level | Up to Week 6
Time course of corrected serum calcium level | Up to Week 6
Time course of calcium-phosphorus product | Up to Week 6
Time course of intact parathyroid hormone | Up to Week 6
Percentage of subjects who achieved the target serum phosphorus level (3.5 to 6.0 mg/dL) | Up to Week 6
Time achievement of the target serum phosphorus level (3.5 to 6.0 mg/dL) | Up to Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (11):
- Japan (11):
  - Site JP00011, Okazaki, Aichi-ken
  - Site JP00009, Chiba, Chiba
  - Site JP00010, Chiba, Chiba
  - Site JP00006, Ibaraki, Ibaraki
  - Site JP00007, Ibaraki, Ibaraki
  - Site JP00008, Ibaraki, Ibaraki
  - Site JP00001, Miyagi, Miyagi
  - Site JP00002, Miyagi, Miyagi
  - Site JP00003, Nagano, Nagano
  - Site JP00004, Nagano, Nagano
  - Site JP00005, Nagano, Nagano

IPD SHARING:
Plan to Share IPD: Undecided